CLINICAL TRIAL: NCT02341898
Title: Implementation of a Multicomponent Intervention to Prevent Physical Restraints in Nursing Home Residents: a Cluster-randomized Controlled Trial
Brief Title: Implementation of a Multicomponent Intervention to Prevent Physical Restraints in Nursing Home Residents (IMPRINT)
Acronym: IMPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Sascha Köpke, Prof. Dr., University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IMPRINT; 01GY1336A (Other Grant/Funding Number: German Federal Ministry of Education and Research); 01GY1336B (Other Grant/Funding Number: German Federal Ministry of Education and Research)
Record Dates: First submitted 2014-12-16; First posted 2015-01-19 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Dementia
Keywords: nursing home care; physical restraints; dementia; implementation research; cluster-randomized controlled trial
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Updated original programme (Experimental): Educational programme for all nurses (90 min. single information session); training and structured support for nominated key nurses (one-day training workshop); provision of printed study material (evidence-based practice guideline; short versions for nurses, legal guardians, and others; information brochures for relatives); supportive material (poster, mugs etc.)
  Interventions: Other: Educational programme for all nurses; Other: Training and structured support for nominated key nurses; Other: Printed study material; Other: Supportive material (poster, mugs etc.)
- Concise updated programme (Experimental): Training and structured support for nominated key nurses (one-day training workshop); nurses' training will be carried out by key nurses as facultative option; key nurses receive an additional train-the-trainer module to apply the educational programme; provision of printed study material (evidence-based practice guideline; short versions for nurses, legal guardians, and others; information brochures for relatives); supportive material (poster, mugs etc.)
  Interventions: Other: Training and structured support for nominated key nurses; Other: Facultative train-the-trainer module for key nurses; Other: Printed study material; Other: Supportive material (poster, mugs etc.)
- Optimized usual care (Active Comparator): Provision of printed study material (evidence-based practice guideline; short versions for nurses, legal guardians, and others; information brochures for relatives) only
  Interventions: Other: Printed study material

INTERVENTIONS:
Other: Educational programme for all nurses
  Arms: Updated original programme
Other: Training and structured support for nominated key nurses
  Arms: Concise updated programme; Updated original programme
Other: Facultative train-the-trainer module for key nurses
  Arms: Concise updated programme
Other: Printed study material
Other: Supportive material (poster, mugs etc.)
  Arms: Concise updated programme; Updated original programme

SUMMARY:
Background: Physical restraints as bedrails and belts are still regularly applied in German nursing homes despite clear evidence showing their lack of effectiveness and safety. In a cluster-randomized controlled trial, the efficacy of a guideline-based multicomponent intervention has been shown with a significant reduction in physical restraints use without adverse events. The present study aims to apply different versions of the original intervention in nursing home residents in four different regions throughout Germany in order to evaluate the effectiveness of the programme.

Methods/Design: Pragmatic cluster-randomized controlled trial comparing two intervention groups ((1) updated original programme and (2) brief version of the updated programme) with a control group (3) receiving printed study materials (optimized usual care). Intervention (1) consists of an information programme for all nurses, additional training and structured support for nominated key nurses, and provision of printed study material and other supportive material. For intervention (2) nurses' training is only optional carried out facultatively by key nurses who have received an additional train-the-trainer module. The control group (3) receives printed study material only. Overall, 120 nursing homes including approximately 10800 residents will be recruited, randomized to one of the three groups and followed up for 12 months. The primary outcome is defined as proportion of residents with at least one physical restraint at 12 months. Physical restraint use will be assessed by direct observation. Secondary outcomes are residents' quality of life as well as safety parameters as i.g. falls and fall-related fractures. Process and cost measures will also be assessed.

ELIGIBILITY:
Cluster level

Inclusion Criteria:

* randomly selected nursing homes in each region; no specific inclusion criteria will be applied

Exclusion Criteria:

* no specific exclusion criteria will be applied

Individual level

Inclusion Criteria:

* all residents within the cluster present on the day of data collection
* all residents newly admitted to clusters during follow-up and present on the day of follow-up data collection

Exclusion Criteria:

* no specific exclusion criteria will be applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10800 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Proportion of residents with at least one physical restraint assessed through direct observation by blinded research assistants | 12 Months

SECONDARY OUTCOMES:
Residents' quality of life (measured by QoL-AD) | 12 Months
  Will be measured by QoL-AD for a randomly selected subgroup of 10% of residents
Falls and fall-related fractures | 12 Months
Costs within trial period (cost parameters related to the implementation of the intervention as well as outcome-related cost parameters) | 12 Months
  For economic evaluation cost parameters related to the implementation of the intervention will be collected as well as outcome-related costparameters; explicit trial-associated will not be taken into account

OTHER OUTCOMES:
Process evaluation | 12 Months
  Different process parameters will be assessed as e.g. relatives' experiences, staff experiences, leaders' experiences and organizational culture

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Köpke, Prof. Dr., Principal Investigator — University of Lübeck
Locations (4):
- Germany (4):
  - Witten/Herdecke University, Witten, North Rhine-Westphalia
  - Martin-Luther-University Halle-Wittenberg, Halle, Saxony-Anhalt
  - University of Lübeck, Lübeck, Schleswig-Holstein
  - University of Hamburg, Hamburg

REFERENCES:
- [Derived] Abraham J, Kupfer R, Behncke A, Berger-Hoger B, Icks A, Haastert B, Meyer G, Kopke S, Mohler R. Implementation of a multicomponent intervention to prevent physical restraints in nursing homes (IMPRINT): A pragmatic cluster randomized controlled trial. Int J Nurs Stud. 2019 Aug;96:27-34. doi: 10.1016/j.ijnurstu.2019.03.017. Epub 2019 Apr 4. PMID 31014546
- [Derived] Abraham J, Mohler R, Henkel A, Kupfer R, Icks A, Dintsios CM, Haastert B, Meyer G, Kopke S. Implementation of a Multicomponent intervention to Prevent Physical Restraints In Nursing home residenTs (IMPRINT): study protocol for a cluster-randomised controlled trial. BMC Geriatr. 2015 Jul 21;15:86. doi: 10.1186/s12877-015-0086-0. PMID 26195247
- See also: project homepage — http://www.leitlinie-fem.de/